CLINICAL TRIAL: NCT01171482
Title: An Open Label, Phase 2 Trial Comparing Sorafenib and 5-fluorouracil/Mitomycin in Hepatocellular Carcinoma With Pulmonary Metastasis
Brief Title: Comparison Study of Sorafenib and 5-fluorouracil/Mitomycin for Metastatic Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There were problems with national reimbursement policies.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-2010-010
Record Dates: First submitted 2010-07-22; First posted 2010-07-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil; Mitomycin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The FM group (Experimental): Patients in the FM group will be administered 5-FU plus mitomycin
  Interventions: Drug: 5-FU; Drug: Mitomycin
- The sorafenib group (Active Comparator): Patients in the sorafenib group will be administered sorafenib
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: 5-FU — 15mg/kg/day continuous IV from day 1 to day 6 every 28 days.
  Other Names: 5-fluorouracil
  Arms: The FM group
Drug: Mitomycin — 4mg/day IV push from day 1 to day 4 every 28 days
  Arms: The FM group
Drug: sorafenib — 400 mg BID every 28 days
  Other Names: Nexavar
  Arms: The sorafenib group

SUMMARY:
The aim of this study is to compare the efficacy of sorafenib to 5-fluorouracil/mitomycin in HCC patients with pulmonary metastasis whose intrahepatic tumors has been controlled with locoregional therapies.

DETAILED DESCRIPTION:
Most HCC patients are diagnosed at advanced stages in Korea, but effective treatment strategies for advanced HCC have not been established. In particular, optimal treatment strategy for extrahepatic as well as intrahepatic recurrences following locoregional therapy (e.g., transarterial chemoembolization, radiofrequency ablation therapy, and percutaneous ethanol injection) is still a challenging issue. Extrahepatic metastasis has been encountered more frequently, being more problematic than before in the management of HCC due to the increased survival with effective locoregional treatments. The lung is the most common site of extrahepatic metastasis and the surgical resection of pulmonary metastatic lesions may result in improved survival in selected patients. Previous studies suggested that aggressive management including resection of the extrahepatic recurrence combined with locoregional therapy for intrahepatic HCC may offer long-term survival in selected patients with recurrent HCC following hepatectomy. Such an aggressive strategy has serious limitation in clinical practice in that extrahepatic recurrence usually present as multiple lesions. Systemic chemotherapy has been one of the most commonly used treatment modalities for patients with multiple extrahepatic metastasis. However, chemotherapy using either a single or combined cytotoxic agents provides only limited benefit for such patients. The aim of this study is to compare the efficacy of sorafenib to 5-fluorouracil/mitomycin in HCC patients with pulmonary metastasis whose intrahepatic tumors had been previously controlled with repeated locoregional therapies before the initiation of systemic chemotherapy.

Outline:

* Experimental arm(the FM group): Patients receive 5-FU IV continuously over 10 hours on day 1~6 and mitomycin IV push on day 1~4. Treatment repeats every 28 days.
* Active Comparator arm(the sorafenib group): Patients will receive 2 tablets of sorafenib (200 mg/tablet) twice daily, orally on a continuous basis.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity. During the treatment period, patients will have study visits on Day 1 of every cycle (every 4 weeks from start of study drug) and will receive CT/MRI assessment every 2 cycles (every 8 weeks). In the event of radiological progression confined to the liver, e.g. appearance of new nodules in the liver in areas previously not treated by locoregional therapies, patients will then also be treated with locoregional therapies such as TACE or local ablation as long as the they may still benefit from treatment. If patients are no longer amenable to locoregional therapies (in the case of untreatable progression), the study will be stopped and best supportive care be offered. This will be based on the investigator's clinical judgment of the subject's status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical or histological diagnosis of HCC based on the guidelines of the AJCC
* Patients with at least one, bi-dimensionally measurable, pulmonary metastasis without intrahepatic viable tumor (Viable tumor is defined as uptake of contrast agent in the arterial phase of dynamic CT or MRI.)
* Patients who have received previous local therapy treatments (RFA, PEI, cryoablation, surgery, resection) to non-target lesions are eligible
* Age : 20 years to 80 years
* ECOG Performance Status of 0 to 1
* Child-Pugh class A or B (Child-Pugh score 7)
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hb ≧ 9 g/dL
  * Absolute neutrophil count > 1000/mm3
  * Platelet count ≧ 60,000 /mm3
  * Adequate clotting function: INR < 1.5
  * Hepatic: AST and ALT < 5 X ULN
  * Renal: serum creatinine < 1.7mg/dL
  * Bilirubin ≦ 3 mg/dL

Exclusion Criteria:

* Patients with diffuse infiltrative type of HCC that are poorly defined
* Presence of hepatic encephalopathy and intractable ascites
* Patients who are on a liver transplant list
* The patient has received prior systemic chemotherapy
* History of organ allograft
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0), including spontaneous bacterial peritonitis
* History of cardiac disease: congestive heart failure > NYHA class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is allowed), cardiac arrhythmias requiring anti-arrhythmic therapy or uncontrolled hypertension and diabetes mellitus
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted
* HIV infection or AIDS-related illness or serious acute or chronic illness (based on medical history)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | every 8 weeks

SECONDARY OUTCOMES:
Time-to-progression (TTP) | every 8 weeks
Objective tumor response rate | Determined by CT scan at the end of every 2 cycles until progressive disease is documented or intolerable toxicity occurs
Adverse event rates and the toxicities | every 4 weeks
Overall survival | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No